CLINICAL TRIAL: NCT05353439
Title: Phase I Dose Escalation and Expansion Study of Tazemetostat in Combination With Topotecan and Pembrolizumab in Recurrent Small Cell Lung Cancer
Brief Title: Testing of Tazemetostat in Combination With Topotecan and Pembrolizumab in Patients With Recurrent Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-03215; NCI-2022-03215 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-C-0005; 10445 (Other: National Cancer Institute LAO); 10445 (Other: CTEP)
Record Dates: First submitted 2022-04-23; First posted 2022-04-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Limited Stage Lung Small Cell Carcinoma; Platinum-Resistant Lung Small Cell Carcinoma; Platinum-Sensitive Lung Small Cell Carcinoma; Recurrent Extensive Stage Lung Small Cell Carcinoma; Recurrent Lung Small Cell Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Biopsy; Specimen Handling; pembrolizumab; tazemetostat; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tazemetostat, pembrolizumab, topotecan) (Experimental): Patients receive tazemetostat PO BID for 7 days prior to cycle 1 and then on days 1-21 of each cycle, pembrolizumab IV over 30 minutes on day 1 of each cycle, and topotecan IV over 30 minutes on days 1-3 or days 1-5 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan throughout the study and undergo biopsy and collection of blood on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab; Drug: Tazemetostat Hydrobromide; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Drug: Tazemetostat Hydrobromide — Given PO
  Other Names: EPZ-6438 Monohydrobromide; Tazemetostat Monohydrobromide; TAZVERIK
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of tazemetostat in combination with topotecan and pembrolizumab in treating patients with small cell lung cancer that has come back after a period of improvement (recurrent). Tazemetostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving tazemetostat in combination with topotecan and pembrolizumab may shrink or stabilize recurrent small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of tazemetostat hydrobromide (tazemetostat) in combination with topotecan hydrochloride (topotecan) and pembrolizumab in patients with recurrent extensive stage (ES)-small cell lung cancer (SCLC), by reviewing dose-limiting toxicities (DLTs) in cycle 1 (21 days). (Dose-Escalation Cohort) II. To select the recommended phase II dose (RP2D) for a combination of tazemetostat, topotecan and pembrolizumab, based on pharmacodynamic (PD) parameters as well as overall efficacy and tolerability. (Dose-Escalation Cohort) III. To evaluate safety and tolerability of tazemetostat in combination with topotecan and pembrolizumab. (Expansion Cohort)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine in a very preliminary fashion, the efficacy of a combination of tazemetostat, topotecan and pembrolizumab in recurrent ES-SCLC by assessing overall response rate (ORR), progression-free survival (PFS), duration of response (DOR) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to ribonucleic acid (RNA) sequencing (RNA-Seq).

II. To assess modulation of EZH2 targets including SLFN11 and MHC among others. III. To identify potential predictive biomarkers of response. IV. To identify mechanisms of drug sensitivity and resistance using deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

V. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

VI. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the Early-Phase and Experimental Clinical Trials Biospecimen Bank (EET Biobank) at Nationwide Children's Hospital.

VII. To characterize circulating cell-free DNA (cfDNA).

OUTLINE: This is a dose-escalation study of tazemetostat followed by a dose-expansion study.

Patients receive tazemetostat orally (PO) twice daily (BID) for 7 days prior to cycle 1 and then on days 1-21 of each cycle, pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle, and topotecan IV over 30 minutes on days 1-3 or days 1-5 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan throughout the study and undergo biopsy and collection of blood on study.

After completion of study treatment, patients are followed every 3 months after removal from study treatment until study closure or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled to the primary cohort must have limited- or extensive-disease SCLC at diagnosis, with relapse at study entry with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, and with prior therapy with platinum doublet. Patients with extensive stage disease should have received chemo-immunotherapy. Both platinum-sensitive and platinum-resistant patients will be included
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of pembrolizumab in combination with tazemetostat and topotecan in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 70%)
* Leukocytes >= 3000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 × ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< 1.5 institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2

  * Note: Creatinine clearance (CrCl) should be calculated per institutional standard. Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated (a)PTT =< 1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load (CD4 count of greater than 250 cells/mcL) within 6 months are eligible for this trial. They must not be receiving prophylactic therapy for an opportunistic infection
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if they are symptomatically stable while off steroid therapy for a minimum of 7 days
* Patients should be class 2B or better on the New York Heart Association Functional Classification
* Ability to understand and the willingness to sign a written informed consent document
* The effects of pembrolizumab and tazemetostat on the developing human fetus are unknown. For this reason and because monoclonal antibodies, EZH2 inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment and for 6 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study treatment administration

Exclusion Criteria:

* Patients who have had chemotherapy, immune checkpoint inhibitors, or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.

  * Note: Patients who have had palliative radiotherapy may be included as long as they have recovered from any radiotherapy related adverse events (allow at least 3 days between radiotherapy completion and study treatment)
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1).

  * Note: Patients with =< grade 2 neuropathy or =< grade 2 alopecia are an exception to this criterion and may qualify for the study
  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Untreated immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI)
* Patients who are receiving any other investigational agents
* Patients with symptomatic brain metastasis are not eligible due to their extremely poor prognosis and since it is unclear whether the investigational agent penetrates the blood-brain barrier. However, subjects who have had treatment for their brain metastasis and are symptomatically stable while off steroid therapy for a minimum of 7 days may be enrolled. The use of physiologic doses of corticosteroids may be approved after consultation with the study PI
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab and tazemetostat or other agents used in study
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients with uncontrolled intercurrent illness but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because pembrolizumab as a monoclonal antibody, and tazemetostat as a EZH2 inhibitor may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab or tazemetostat, breastfeeding should be discontinued if the mother is treated with these agents and for 1 week after the last dose of tazemetostat. These potential risks may also apply to other agents used in this study
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C
* Has received a live vaccine within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted
* Has thrombocytopenia, neutropenia, or anemia of grade >= 3 (per Common Terminology Criteria for Adverse Events [CTCAE] 5.0 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)
* Has abnormalities known to be associated with MDS (e.g. del 5q, chromosome [chr] 7 abnormality [abn]) and myeloproliferative neoplasm (MPN) (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing
* Has a prior history of T-cell lymphoblastic lymphoma (T-LBL), T-cell acute leukemia (T-ALL) or B-cell acute lymphoblastic leukemia (B-ALL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (dose-escalation cohort) | Up to 21 days (cycle 1)
Incidence of adverse events (expansion cohort) | Up to 3 years
  Will be evaluated in more detail by reporting the adverse events noted, by type and grade, for the patients in the expansion cohort.

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years
  Will be estimated based on patients evaluable for response and will be presented along with a 95% confidence interval.
Progression-free survival | From the on-study date until the date of progression or death without progression, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method, resulting in median survival times with 95% confidence interval.
Overall survival | From the on-study date until the date of death or last follow-up, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method, resulting in median survival times with 95% confidence interval.
Duration of response | From the first date of response to the date of progression, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method, resulting in median survival times with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, Principal Investigator — National Cancer Institute LAO
Locations (15):
- United States (15):
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm